CLINICAL TRIAL: NCT01790945
Title: Diabetic Macular Edema and Diabetic Retinopathy Identification by Screening (Telemed) With Verified Automated Retinal Photography
Brief Title: Diabetic Macular Edema and Diabetic Retinopathy Screening (TeleMed) With Automated Retinal Photography
Acronym: DIVER
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Retina Institute of Hawaii (Other)
Responsible Party: Sponsor
Other Study IDs: DIVER Study
Record Dates: First submitted 2013-02-11; First posted 2013-02-13 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Mild Nonproliferative Diabetic Retinopathy; Moderate Nonproliferative Diabetic Retinopathy; Severe Nonproliferative Diabetic Retinopathy; Proliferative Diabetic Retinopathy; Diabetic Macular Edema

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment Study: Population of subjects will have been diagnosed with mild NPDR, Moderate NPDR, Severe NPDR, PDR and DME

SUMMARY:
The purpose of this study is explore if a partnership and screening program put in place between a busy retina practice and their referring diabetes care offices can improve diabetic retinopathy and diabetic macular edema diagnosis, care and overall diabetes control in patients with diabetic eye disease.

DETAILED DESCRIPTION:
Retina Institute of Hawaii will place an infrastructure to screen for diabetic retinopathy/diabetic macular edema in 5 of the states largest Primary Care Clinics, General Medical and or Endocrine practices which re our primary referrals for diabetes patients. Each Sub-site will receive a DRS Automated Retinal Camera and our staff will train the sub-site's staff on taking images. The submission of these images to our practice will be administered by an automated job scheduler in the DRS Automated Retinal Camera removing the requirement of the locations to send images. Images will be electronically uploaded and sent to the Retina Institute of Hawaii for detailed interpretation and report sent back to the patients, their diabetes care MD's and their nurse practitioners/diabetic educators.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with diabetes that have not seen an Ophthalmologist in the past 1 year

Exclusion Criteria:

* Patients with diabetes already under the care of an Ophthalmologist.
* Patient not willing to give Consent for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: (n=500) A large population will need to be screened to find 100-150 patients with diabetic eye disease
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-06 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
% change in Diabetic Retinopahy/Diabetic Macular Edema diagnosis with pre-screening system compared to post-screening system | 6 months

SECONDARY OUTCOMES:
Change in HgA1C from Primary Care Physician referral to post retinal specialist visit | six months

OTHER OUTCOMES:
Time from PCP referral for patient to see an ophthalmologist and appointment with retinal specialist | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Bennett, MD, Principal Investigator — Retina Institute of Hawaii
Locations (1):
- Craig Kadooka, MD, Hilo, Hawaii, United States